CLINICAL TRIAL: NCT06360939
Title: Radiotherapy vs Catheter Ablation for Ventricular Tachycardia in Structural Heart Disease
Acronym: Radioablate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Collaborators: University of Sydney (Other); National Heart Foundation, Australia (Other)
Responsible Party: Principal Investigator, Saurabh Kumar, Associate Professor, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETH02659
Record Dates: First submitted 2024-01-02; First posted 2024-04-11 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Tachycardia; Cardiomyopathies; Arrhythmias, Cardiac; Ventricular Arrythmia
Keywords: catheter ablation; stereotactic body radiation therapy; non invasive; radioablation
MeSH Terms: conditions — Tachycardia, Ventricular; Cardiomyopathies; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic body radiation therapy (Experimental): SBRT within 6 weeks of randomisation guided by previous electrophysiology studies, electrocardiograms and cardiac imaging.
  Interventions: Radiation: SBRT
- Catheter ablation (Active Comparator): CA within 6 weeks of randomisation (constituting standard of care for patients with VT and structural heart disease)
  Interventions: Procedure: CA

INTERVENTIONS:
Radiation: SBRT — Delivery of 25Gy in a single dose fraction to target area within 6 weeks of randomization
  Arms: Stereotactic body radiation therapy
Procedure: CA — CA (endocardial and/or epicardial at operator discretion) within 6 weeks of randomization.
  Arms: Catheter ablation

SUMMARY:
The goal of this randomized clinical trial is to test the efficacy of stereotactic body radiation therapy (SBRT) in treating ventricular tachycardia (VT) in patients with advanced structural heart disease. The main questions it aims to answer are:

* What is the efficacy of SBRT compared to catheter ablation (CA) in achieving a ≥ 75% reduction in VT burden at 6 months
* What is the comparable safety profile of SBRT vs CA Researchers will compare SBRT and CA (standard of care).

DETAILED DESCRIPTION:
Hypothesis

We hypothesise that in an open label randomised controlled trial of patients with advanced structural heart disease and ventricular tachycardia (VT) that stereotactic body radiation therapy (SBRT) will be superior in reducing VT burden compared to standard care comprising of catheter ablation (CA) and routine medical care with acceptable safety and adverse events.

Aims

This is a trial to examine if in an open label randomised trial of 60 patients with structural heart disease and VT followed for 3 years with a minimum follow up of 1 year of SBRT compared CA results in:

1. An improvement in a primary outcome of proportion of patients with a ≥75% reduction in VT burden in the 6 months following intervention compared to the 6 months intervention
2. Comparable safety profile (serious adverse events [SAE] and adverse events of special interest [AESI] at 6 months;
3. reduction in secondary endpoints at 6, 12, 24 and 36 months of: any VT recurrence, absolute % reduction in VT burden compared to 6 months pre-treatment, number of anti-arrhythmic drugs (AADs) compared to pre-treatment, cardiovascular hospitalisation, all-cause mortality, cardiac transplantation, combined endpoint of cardiovascular hospitalisation/transplant/mortality, SAE and AESI from treatment, ventricular function abd change of quality of life (QOL) metrics (at 12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Structural heart disease (including ischaemic cardiomyopathy , non-ischaemic cardiomyopathy or congenital heart disease and defined as any one of

   1. segmental or global decreased ventricular wall motion as defined by TTE, CT or cMRI
   2. myocardial hypertrophy
   3. myocardial scar (evidenced by late gadolinium enhancement on cMRI, wall thinning on cardiac CT, low voltage on electrophysiological study or abnormal intracardiac echocardiography)
2. Recurrent monomorphic VT which can include

   1. at least one episode of VT treated by ICD and/or
   2. sustained VT (lasting >30s) and/or
   3. inducible sustained VT on invasive electrophysiological study (EPS) or non-invasive programmed stimulation (NIPS)
3. PAINESD score of ≥9 points and/or at least moderate risk of VT recurrence or death as defined by the I-VT score. Both are validated tools used clinically to identify patient at high risk of VT recurrence and/or mortality after CA.

Exclusion Criteria:

1. Age < 18 years
2. Life expectancy < 3 months
3. Catheter ablation deemed futile or with prohibitive risk by cardiac electrophysiologist.
4. Unwilling or unable to provide consent
5. Known cardiac channelopathies (e.g. Catecholaminergic polymorphic ventricular tachycardia (CPVT), long- or short QT syndrome, Brugada syndrome)
6. Contraindications to radiotherapy as deemed by referring physician and/or radiation oncologist
7. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
VT burden | 6 months
  Change in proportion of patients with a ≥75% reduction in VT burden at 6 months (number of VT episodes in 6 months post treatment compared to the number of VT episodes in the 6 months prior to randomisation excluding a 6-week blanking period after treatment initiation)

SECONDARY OUTCOMES:
Recurrent sustained VT | 6, 12, 24 and 36 months
  Recurrent sustained VT ascertained by implanted cardioverter defibrillator (ICD) (VT identified and treated by the ICD with anti-tachycardia pacing (ATP) and/or internal ICD delivered shock or ≥30 seconds of VT if untreated by ICD
VT storm | 6, 12, 24 and 36 months
  VT storm (three or more documented episodes of VT within 24 hours or incessant VT)
Absolute VT burden | 6, 12, 24 and 36 months
  Absolute percentage reduction in VT burden compared to pre-ablation
Serious Adverse Events (SAE) and Adverse Events of Special Interest (AESI) | At all time points up to 36 months
  1. SAE and AESI related to effects of SBRT
  2. SAE and AESI related to standard care e.g. medical anti-arrhythmic drug therapy or catheter ablation or heart transplantation
ICD shocks | 6, 12, 24 and 36 months
  Implantable Cardioverter Defibrillator shocks
Hospitalization | 6, 12, 24 and 36 months
  Cardiovascular as well as specifically heart failure and arrhythmia
All cause mortality | 6,12, 24 and 36 months
  All cause mortality
Cardiovascular Mortality | 6,12, 24 and 36 months
  Cardiovascular mortality
Composite outcome of VT recurrence/hospitalisation/death/ cardiac transplantation | 6,12, 24 and 36 months
  Composite outcome as above
Ventricular function | 6,12, 24 and 36 months
  As determined by echocardiography (ejection fraction, speckle tracking echocardiography)
Quality of Life as per Short Form - 36 (SF-36) Score | 6,12, 24 and 36 months
  Change in quality of life at 6 and 12 months (compared to pre-intervention) as measured by Short Form- 36 (SF-36) [0-100 scale, 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability].
Quality of Life as per Implantable Cardioverter Defibrillator Concerns Questionnaire (ICDC) score | 6,12, 24 and 36 months
  Change in quality of life at 6 and 12 months (compared to pre-intervention) as measured by Implantable Cardioverter Defibrillator Concerns Questionnaire (ICDC) score. [0-100 scale, 100 equivalent to maximum concern]
Number of AADs | 6,12, 24 and 36 months
  Number of AADs at time points following randomization

IPD SHARING:
Plan to Share IPD: No